CLINICAL TRIAL: NCT07401524
Title: Carbetocin Administration for the Prevention of Postpartum Hemorrhage in Twin Deliveries: A Randomized Controlled Trial
Brief Title: Carbetocin Uterotonic Treatment in Twin Pregnancies for Prevention of Postpartum Hemorrhage
Acronym: CUTT-PPH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Avihu Krieger, Principal Investigator and Physician, Department of Obstetrics and Gynecology, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMC-26-2925
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Hemorrhage; Twin Pregnancy
Keywords: Carbetocin; Oxytocin; Twin Delivery; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Intervention Model Description: Parallel-group, single-center randomized controlled trial with 1:1 allocation comparing prophylactic carbetocin versus standard oxytocin administered immediately after delivery of the second twin (vaginal or cesarean).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin (Experimental): Participants in this arm will receive a single intravenous dose of carbetocin immediately after delivery of the second twin, as prophylaxis for postpartum hemorrhage, following either vaginal or cesarean delivery.
  Interventions: Drug: Carbetocin
- Oxytocin (Standard Care) (Active Comparator): Participants in this arm will receive standard prophylactic oxytocin according to institutional protocol, following either vaginal or cesarean delivery.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin will be administered as a single intravenous dose immediately following delivery of the second twin, according to institutional protocol, for the prevention of postpartum hemorrhage.
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin will be administered intravenously according to standard institutional practice, for the prevention of postpartum hemorrhage.
  Arms: Oxytocin (Standard Care)

SUMMARY:
The goal of this clinical trial is to learn if the drug carbetocin works better than standard care to prevent heavy bleeding after childbirth in people carrying twin pregnancies. Heavy bleeding after delivery, also called postpartum hemorrhage, is more common after twin births and can lead to anemia, blood transfusions, and other serious health problems.

In this study, bleeding will be evaluated by measuring how much blood hemoglobin levels drop from before delivery to the day after delivery.

The main questions this study aims to answer are:

* Does giving carbetocin after delivery lower blood loss compared with standard oxytocin treatment?
* Is carbetocin safe and practical to use in twin deliveries?

Researchers will compare carbetocin to standard oxytocin treatment to see which approach better prevents bleeding after twin vaginal or cesarean delivery.

Participants will:

* Be randomly assigned to receive either carbetocin or standard oxytocin after the second twin is delivered
* Have blood tests before delivery and on the day after delivery
* Be followed during their hospital stay and for up to six weeks after delivery for safety outcomes

DETAILED DESCRIPTION:
Postpartum hemorrhage is a major cause of maternal morbidity worldwide and occurs more frequently in twin pregnancies compared with singleton deliveries. Uterine overdistension in multiple gestations increases the risk of uterine atony, the leading cause of postpartum hemorrhage. Preventive uterotonic therapy is therefore a central component of routine care following twin delivery.

Carbetocin is a long-acting synthetic analogue of oxytocin that induces sustained uterine contraction and is approved for the prevention of postpartum hemorrhage. Previous randomized trials and meta-analyses have demonstrated that carbetocin is associated with reduced need for additional uterotonic agents and blood transfusion compared with oxytocin, primarily in cesarean deliveries. However, data specific to twin pregnancies are limited, and no randomized controlled trial has directly compared carbetocin with standard oxytocin prophylaxis in a twin population including both vaginal and cesarean deliveries.

This single-center randomized controlled trial is designed to evaluate the effectiveness and safety of prophylactic carbetocin compared with standard oxytocin for the prevention of postpartum hemorrhage in twin deliveries. Pregnant individuals aged 18 years or older with twin pregnancies delivering at or beyond 23 weeks of gestation will be eligible to participate. Following written informed consent, participants will be randomized in a 1:1 ratio to receive either carbetocin or standard oxytocin immediately after delivery of the second twin.

Randomization will be performed using computer-generated permuted block sequences to ensure balanced group allocation. The assigned uterotonic treatment will be administered according to group assignment as part of routine postpartum care. Participants in the intervention group will receive a single intravenous dose of carbetocin, while participants in the control group will receive intravenous oxytocin according to institutional protocol.

Maternal hemoglobin levels will be obtained as part of routine clinical care prior to delivery and again on the first postpartum day. The primary outcome of the study is the change in maternal hemoglobin from before delivery to postpartum day one, serving as an objective measure of postpartum blood loss. Secondary outcomes include estimated blood loss, clinical postpartum hemorrhage, need for additional uterotonic agents, blood product transfusion, use of additional medical or surgical interventions for bleeding, maternal infections, intensive care unit admission, and length of postpartum hospitalization.

Participants will be followed throughout their delivery hospitalization and for up to six weeks postpartum to assess maternal outcomes and safety. Adverse events will be monitored by the clinical care team and reviewed in accordance with institutional policies. All data will be collected from the electronic medical record and stored in a secure, password-protected research database using unique study identifiers to maintain confidentiality.

The planned sample size is 120 participants, which is expected to provide sufficient power to detect a clinically meaningful difference in postpartum hemoglobin change between groups while ensuring adequate representation of both vaginal and cesarean deliveries. This trial aims to provide high-quality evidence regarding the role of carbetocin in preventing postpartum hemorrhage in twin pregnancies and to inform future clinical practice in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals aged ≥18 years
* Twin pregnancies
* Gestational age ≥23 weeks

Exclusion Criteria:

* Known hypersensitivity or contraindication to carbetocin
* Higher-order multiple gestation (triplets or more)
* Maternal age <18 years
* Known placenta accreta spectrum
* Known bleeding disorder
* Intrauterine fetal death of one or more fetuses
* Hyponatremia precluding oxytocin use
* Planned delivery at a non-participating hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in maternal hemoglobin level from baseline to postpartum | The most recent hemoglobin measurement taken within 30 days prior to delivery to the day after delivery.
  The primary outcome is the change in maternal hemoglobin level, defined as the difference between pre-delivery hemoglobin and hemoglobin measured on the day after delivery.

SECONDARY OUTCOMES:
Estimated Blood Loss Measured by Quantitative Clinical Assessment | During delivery (vaginal delivery or cesarean delivery)
  Estimated blood loss during delivery, assessed using standard quantitative clinical methods as documented in the medical record.
Number of Participants With Early Postpartum Hemorrhage | From delivery up to 24 hours postpartum.
  Early postpartum hemorrhage defined as quantitative blood loss >500 mL after vaginal delivery or >1000 mL after cesarean delivery.
Number of Participants With Late Postpartum Hemorrhage | From 24 hours postpartum up to 6 weeks postpartum.
  Late postpartum hemorrhage defined as quantitative blood loss >500 mL after vaginal delivery or >1000 mL after cesarean delivery.
Number of Participants Requiring Additional Uterotonic Administration | From delivery up to 6 weeks postpartum
Number of Participants Receiving Tranexamic Acid | From delivery up to 6 weeks postpartum
Number of Participants Receiving Blood Product Transfusion | From delivery up to 6 weeks postpartum.
Number of Blood Products Transfused | From delivery up to 6 weeks postpartum.
Post delivery day 1 hemoglobin level. | Post delivery day 1
Number of Participants Requiring Intrauterine Balloon Tamponade | From delivery up to 6 weeks postpartum
Use of uterine compression sutures (e.g., B-Lynch suture). | From delivery up to 6 weeks postpartum.
Number of Participants Undergoing Hysterectomy | From delivery up to 6 weeks postpartum.
Number of Participants Admitted to the Intensive Care Unit | From delivery up to 6 weeks postpartum.
  Admission to an intensive care unit for maternal indications as documented in the medical record.
Number of Participants With Maternal Postpartum Infections | From delivery up to 6 weeks postpartum.
  Includes postpartum fever, endometritis, urinary tract infection, mastitis, and surgical site infection.
Maternal death. | From delivery up to 6 weeks postpartum.
Length of postpartum hospitalization. | From delivery up to 6 weeks postpartum
Number of Participants Re-admitted Within 6 Weeks Postpartum Due to Bleeding | From delivery up to 6 weeks postpartum.
Number of Participants Requiring Additional Surgical Intervention Within 6 Weeks Postpartum | From delivery up to 6 weeks postpartum.
Number of Participants Breastfeeding at 6 Weeks Postpartum | 6 weeks postpartum.
Side effects and adverse outcomes | From delivery up to 24 hours postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
This study is planned as a single-center trial, and at this stage, there are no plans or agreements in place for sharing individual participant data (IPD). Future considerations for data-sharing agreements may be evaluated based on future research collaborations and institutional policies.